CLINICAL TRIAL: NCT04513704
Title: Oral Semaglutide Pharmacokinetics in Healthy Subjects, Effect of Dosing Schedules
Brief Title: A Clinical Trial Comparing Semaglutide in Healthy People Who Eat and Take the Medicine at Different Times
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-4556; U1111-1243-9641 (Other: World Health Organization (WHO)); 2019-004569-42 (Registry Identifier: European Medicines Agency (EudraCT))
Record Dates: First submitted 2020-08-12; First posted 2020-08-14 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Healthy Volunteers Type 2 Diabetes
MeSH Terms: interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Oral Semaglutide A (Experimental): Participants will receive oral semaglutide tablet once daily for 10 days (3 mg for first 5 days and 7 mg for the next 5 days), with a pre-specified timing for 2 hours of the pre-dose fast, followed by a 30 minutes post-dose fast.
  Interventions: Drug: Oral Semaglutide
- Oral Semaglutide B (Experimental): Participants will receive oral semaglutide tablet once daily for 10 days (3 mg for first 5 days and 7 mg for the next 5 days), with a pre-specified timing for 4 hours of the pre-dose fast, followed by a 30 minutes post-dose fast.
  Interventions: Drug: Oral Semaglutide
- Oral Semaglutide C (Experimental): Participants will receive oral semaglutide tablet once daily for 10 days (3 mg for first 5 days and 7 mg for the next 5 days), with a pre-specified timing for 6 hours of the pre-dose fast, followed by a 30 minutes post-dose fast.
  Interventions: Drug: Oral Semaglutide
- Oral Semaglutide D (Experimental): Participants will receive oral semaglutide tablet once daily for 10 days (3 mg for first 5 days and 7 mg for the next 5 days), with a pre-dose fasting time of 2 hours followed by a post-dose overnight fast.
  Interventions: Drug: Oral Semaglutide
- Oral Semaglutide E (Active Comparator): Participants will receive oral semaglutide tablet once daily for 10 days (3 mg for first 5 days and 7 mg for the next 5 days). Participants will be instructed to take the trial product in the morning after an overnight fast and wait 30 minutes before taking any food, water or other oral medication in accordance with the approved dosing schedule for oral semaglutide.
  Interventions: Drug: Oral Semaglutide

INTERVENTIONS:
Drug: Oral Semaglutide — Participants will receive oral semaglutide tablet once daily for 10 days (3 mg for first 5 days and 7 mg for the next 5 days).

SUMMARY:
The goal of this trial is to find out whether taking semaglutide tablets at different times before and after eating has a similar effect compared to the recommended dosing time. Participants with type 2 diabetes are recommended to take semaglutide on an empty stomach, and they should not eat, drink, or take any oral medicine for at least 30 minutes after that. The trial will look at how different dosing times of semaglutide before and after eating a meal changes how much semaglutide participants get into their blood. Participants will get one semaglutide tablet daily for a total of 10 days. For the first 5 days participants will receive semaglutide tablets of 3 mg and for the next 5 days, participants will receive semaglutide tablets of 7 mg. From here onwards, semaglutide tablets will be referred to as the 'trial medicine', unless specifically mentioned. Participants will get the trial medicine (3 mg and 7 mg) under one of the 5 following dosing conditions. It will be decided by chance under which dosing condition participants will receive the trial medicine: A 2 hour fast before taking the trial medicine and 30 minutes fast after taking the trial medicine (Test arm A), A 4 hour fast before taking the trial medicine and 30 minutes fast after taking the trial medicine (Test arm B), A 6 hour fast before taking the trial medicine and 30 minutes fast after taking the trial medicine (Test arm C), A 2 hour fast before taking the trial medicine and an overnight fast (at least 6 hours fast) after taking the trial medicine (Test arm D), An overnight fast before taking the trial medicine and 30 minutes fast after taking the trial medicine (Reference arm E). Before each fasting period prior to receiving the trial medicine, participants will fast for 4 hours and then receive a standardised meal. The meal should be completed before the 2, 4 or 6 hours fasting is started. The trial will last for about 48 to 78 days (about 1.5 to 2.5 months). Participants will have 4 scheduled visits with the study doctor. At one of the visits, participants will be admitted to the trial unit and have to stay for 12 consecutive days. At all visits participants will meet with trial staff and will have blood tests along with other clinical checks and tests. Participants will be asked about their health, medical history, and habits. Women only: Women cannot take part if pregnant, breast-feeding, or planning to become pregnant during the trial period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18-64 years (both inclusive) at time of signing informed consent.
* Body mass index (BMI) between 20.0 and 29.9 kg/m^2 (both inclusive).
* Considered to be generally healthy based on the medical history, physical examination, and the results of vital signs, electrocardiogram and clinical laboratory tests performed during the screening visit, as judged by the investigator.

Exclusion Criteria:

* Glycated haemoglobin (HbA1c) greater than or equal to 6.5% (48 mmol/mol) at screening.
* Use of tobacco and nicotine products, defined as any of the below:

  * Smoking more than 5 cigarettes or the equivalent per day
  * Not willing to refrain from smoking and use of nicotine substitute products during the in-house period.
* Presence of clinically significant gastrointestinal disorders or symptoms of gastrointestinal disorders potentially affecting absorption of drugs or nutrients, as judged by the investigator.
* Personal or first-degree relative(s) history of multiple endocrine neoplasia type 2 or medullary thyroid carcinoma (as declared by subject or reported in the medical records).
* Presence or history (as declared by subject or reported in the medical records) of pancreatitis (acute or chronic).
* History (as declared by subject or reported in the medical records) of major surgical procedures involving the stomach potentially affecting absorption of trial products (e.g. subtotal and total gastrectomy, sleeve gastrectomy, gastric bypass surgery).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 156 (Actual)
Dates: Start 2020-08-28 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Area under the semaglutide plasma concentration - time curve during a dosing interval after the 10th dosing (AUC0-24h,sema,day10) | From 0 to 24 hours after the 10th dosing (day 10)
  nmol*h/L

SECONDARY OUTCOMES:
Maximum observed semaglutide plasma concentration after the 10th dosing (Cmax,0-24h,sema,day10) | From 0 to 24 hours after the 10th dosing (day 10)
  nmol/L
Time to maximum observed semaglutide plasma concentration after the 10th dosing (tmax,0-24h,sema,day10) | From 0 to 24 hours after the 10th dosing (day 10)
  hours (h)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure 1452, Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Harrow, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com

REFERENCES:
- [Derived] van Hout M, Forte P, Jensen TB, Boschini C, Baekdal TA. Effect of Various Dosing Schedules on the Pharmacokinetics of Oral Semaglutide: A Randomised Trial in Healthy Subjects. Clin Pharmacokinet. 2023 Apr;62(4):635-644. doi: 10.1007/s40262-023-01223-9. Epub 2023 Mar 17. PMID 36932262